CLINICAL TRIAL: NCT01893671
Title: Observational Study of Corneal Power, Astigmatism, and Aberration Changes After LASIK
Brief Title: Corneal Power, Astigmatism, and Aberration Changes After LASIK
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Professor of Ophthalmology, Oregon Health & Science University, Oregon Health and Science University
Other Study IDs: OHSU IRB#6612; R01EY018184 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Measurements of Patients Using OCT Before and After LASIK
Keywords: LASIK; corneal power; astigmatism; HOA; Optical Coherence Tomography
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LASIK: Subjects undergoing routine LASIK for the correction of myopia or hyperopia.

SUMMARY:
The primary goal of the study is to determine if Optical Coherence Tomography (OCT) measurement of corneal power and astigmatism is more accurate than conventional Placido-ring corneal topography. A second goal is to evaluate OCT-based epithelial thickness mapping. The postoperative epithelial thickness variation will be used to calculate refractive effects and calibrate the smoothing parameter in the mathematical model relating corneal mean curvature and epithelial thickness. A third goal is to assess the repeatability of OCT measurements. A fourth goal is to develop a method of estimating the focusing power, astigmatism, and HOA of the crystalline lens based on measurements of the lens' anterior and posterior capsular topographies and positions with the ultrahigh-speed MIT OCT prototype.

DETAILED DESCRIPTION:
A prospective observational study on refraction and HOA changes after LASIK will be conducted at OHSU and Baylor. We will enroll 50 subjects undergoing routine LASIK for the correction of myopia or hyperopia. The Optovue anterior segment OCT prototype will be used to measure corneal power, astigmatism, HOA, and epithelial thickness map. The ultrahigh-speed MIT OCT prototypes will also be used when they become available. A comprehensive eye examination will be performed preoperatively. OCT scan, manifest refraction, visual acuity, Placido-ring corneal topography, slit scanning/Scheimpflug camera, and wavefront measurements will be acquired preoperatively and 3-6 months after the surgery. The LASIK-induced refraction and wavefront HOA changes will be used as the reference standard to evaluate the accuracy of OCT-measured corneal power, astigmatism, and HOA changes. The primary goal of the study is to determine if OCT measurement of corneal power and astigmatism is more accurate than conventional Placido-ring corneal topography. A second goal is to evaluate OCT-based epithelial thickness mapping. The postoperative epithelial thickness variation will be used to calculate refractive effects and calibrate the smoothing parameter in the mathematical model relating corneal mean curvature and epithelial thickness. A third goal is to assess the repeatability of OCT measurements. A fourth goal is to develop a method of estimating the focusing power, astigmatism, and HOA of the crystalline lens based on measurements of the lens' anterior and posterior capsular topographies and positions with the ultrahigh-speed MIT OCT prototype. The reference standard for lens focusing power and astigmatism will be based on a Gaussian optics model that takes as inputs manifest refraction, crystalline lens position, axial eye length, and OCT corneal power and astigmatism measurements. The reference standard for lens HOA will be the difference between wavefront HOA and corneal HOA. For each eye, the best-fit effective index of the lens will be found so that OCT measurements will match the reference data. Although the lens index is likely to be higher centrally than peripherally, this secondary perturbation will be accounted for by a posterior shift of the posterior lens capsule in OCT images, due to the fact that apparent distances in OCT images is a product of physical distance and optical group index. Thus HOA due to index variation in the lens would translate to unevenness in the posterior capsule surface that could be measured with OCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who qualify for primary LASIK for either myopia or hyperopia, with or without astigmatism.

Exclusion Criteria:

1. Inability to give informed consent.
2. Inability to maintain stable fixation for OCT imaging.
3. Inability to commit to required visits to complete the study.
4. Eyes with concurrent cataract, retinal diseases, glaucoma, or other eye conditions that may limit the visual outcome after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing routine LASIK for the correction of myopia or hyperopia with or without astigmatism
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
OCT measurement of corneal power and astigmatism vs Placido-ring | 5 year
  primary goal of the study is to determine if OCT measurement of corneal power and astigmatism is more accurate than conventional Placido-ring corneal topography

SECONDARY OUTCOMES:
An evaluation of OCT-based epithelial thickness mapping | 5 year
  The postoperative epithelial thickness variation will be used to calculate refractive effects and calibrate the smoothing parameter in the mathematical model relating corneal mean curvature and epithelial thickness.
OCT measurements repeatability | 5 year
  An assessment of the repeatability of OCT measurements
The Development of a method of estimating the focusing power, astigmatism, and HOA of the crystalline lens | 5 year
  The Development of a method of estimating the focusing power, astigmatism, and HOA of the crystalline lens based on measurements of the lens' anterior and posterior capsular topographies and positions with the ultrahigh-speed MIT OCT prototype.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health & Science Universtiy
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States